CLINICAL TRIAL: NCT01967524
Title: Multicenter Randomized Double-blind Study Evaluating the Effects of Botulinum Toxin A Associated With ropivacaïne Versus ropivacaïne Alone in the Treatment of the Myofascial Pelviperineal Pain
Acronym: MYOTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC13_0061
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Myofascial Pelviperineal Pain
Keywords: Myofascial pain; Perineal pain; Chronic pelvic pain; Botulinum toxin type A; Ropivacaïne
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- botulinum toxin A + ropivacaïne (Experimental)
  Interventions: Drug: botulinum toxin A + ropivacaïne
- Ropivacaïne (Active Comparator)
  Interventions: Drug: Ropivacaïne

INTERVENTIONS:
Drug: botulinum toxin A + ropivacaïne — D0 :
  * Calcul of the average of EN (digital scale) (EN completed from D-8 to D-1)
  * QDSA (Saint-Antoine pain questionnaire)
  * QCD (Pain questionnaire)
  * MPI (Multidimensional Pain Inventory)
  * Beck scale
  * HAD (Hospital Anxiety and Depression scale)
  * SF36 (Short Form 36)
  * injection of botulinum toxin A associated with ropivacaïne
  D30, D90, D120 and D150 (phone call): Calcul of the average of EN
  D60 and D180 (on site visits): adverse events reporting, calcul of the average of EN, PGI-I (Patient Global Impression of Improvement), questionnaires (QDSA, QCD, MPI, treatment satisfaction, Beck scale, HAD and SF36).
  Arms: botulinum toxin A + ropivacaïne
Drug: Ropivacaïne — D0 :
  * Calcul of the average of EN (digital scale) (EN completed from D-8 to D-1)
  * QDSA (Saint-Antoine pain questionnaire)
  * QCD (Pain Questionnaire)
  * MPI (Multidimensional Pain Inventory)
  * Beck scale
  * HAD (Hospital Anxiety and Depression scale)
  * SF36 (Short Form 36)
  * injection of ropivacaïne alone
  D30, D90, D120 and D150 (phone call): Calcul of the average of EN
  D60 and D180 (on site visits): adverse events reporting, calcul of the average of EN, PGI-I (Patient Global Impression of Improvement), questionnaires (QDSA, QCD, MPI, treatment satisfaction, Beck scale, HAD and SF36).
  Arms: Ropivacaïne

SUMMARY:
Myofascial pains are frequently found during the clinical examination of the patients presenting a painful chronic syndrome of the pelvis or the perineum. If the physiopathology of this component of the pain characterized by triggerpoints found in the clinical examination, remains uncertain; its coverage contributes to the improvement of the global pain of the patient. The physiotherapy can be useful but when it is not useful, we proposed injections of triggerpoints by local anesthetics. The injections of botulinum toxin on these triggerpoints have a legitimacy (action on the muscular cramp and action on the afferent fibers) but are they superior to the injections of local anesthetics of triggerpoints? The literature remains poor on the subject, justifying this randomized double-blind protocol comparing the efficacy of the botulinum toxin associated with a local anesthetic versus local anesthetic alone with a main criterion of evaluation in 2 months and a monthly follow-up as long as the patient remains improved and maximum in 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient presenting a "dysfunctional" pain of the pelvis or the perineum (without lesional pathology justifying a specific treatment) by an endopelvic touch
* Pain evolving since at least 6 months and persisting in spite of the analgesic treatments and the physiotherapy
* Patient presenting to the clinical examination one or several active triggerpoints found on the internal obturating muscles and/or elevators of the anus, with a maximum of 10 triggerpoints on the whole body.
* Patient presenting an average of the maximal pains of the week before the inclusion superior or equal to 4 and inferior or equal to 9/10 (evaluation of the daily maximal pain on a digital scale from 0 to 10)
* Signed informed consent
* Subjects affiliated with an appropriate social security system

Exclusion Criteria:

* Patients with bleeding risk and anticoagulant therapy
* Intolerance of botulinum toxin A, ropivacaïne and nitrous oxide
* Injection of botulinum toxin in any place whatsoever in the previous 3 months
* Pregnancy and breast feeding
* Antibiotic treatment by aminoglycosides
* Recent anti-inflammatory treatment
* Severe myasthenia
* Lambert-Eaton syndrome
* Patients with neurological disorders, dysphagia, food choking or inhalation pneumonia
* Beck score > 16
* Patients having an average of the maximal pains of the previous week lower than 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evolution of the PGI-I (Patient Global Impression of Improvement) | 2 month
  The main objective is to evaluate the efficacy of injection of botulinum toxin A associated with ropivacaïne versus ropivacaïne alone on the global suffering of chronic myofascial pelviperineal syndromes two month after the injection.
  The success will be defined as an improvement of the PGI-I corresponding to the first 2 levels.

SECONDARY OUTCOMES:
Evaluation of pain on digital scale (EN) | 6 month
  Evaluation of pain on digital scale (EN), each month after the injection
To assess the changing parameters of quality of life: global improvement score / treatment satisfaction assessed by digital scale, international pain scales (MPI, QDSA, QCD) / Beck and HAD score | 6 month
To assess the evolution of analgesics consumption (score MQS) | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques LABAT, Dr, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - Clinique Axium, Aix-en-Provence
  - Besançon University Hospital, Besançon
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - La Réunion University Hospital, Saint Denis de La Réunion

REFERENCES:
- [Derived] Levesque A, Ploteau S, Michel F, Siproudhis L, Bautrant E, Eggermont J, Rabischong B, Volteau C, Perrouin-Verbe MA, Labat JJ. Botulinum toxin infiltrations versus local anaesthetic infiltrations in pelvic floor myofascial pain: Multicentre, randomized, double-blind study. Ann Phys Rehabil Med. 2021 Jan;64(1):101354. doi: 10.1016/j.rehab.2019.12.009. Epub 2020 Jan 22. PMID 31981833